CLINICAL TRIAL: NCT02616731
Title: Oral Tranexamic Acid Versus Diosmin for Treatment of Menorrhagia in Women Using Copper IUD: Randomized Controlled Trial
Brief Title: Oral Tranexamic Acid Versus Diosmin for Treatment of Menorrhagia in Women Using Copper IUD
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ahmed Alanwar, lecturer, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TXAvsDiosmin-IUDmenorrhagia
Record Dates: First submitted 2015-11-22; First posted 2015-11-30 (Estimated); Last update posted 2015-11-30 (Estimated); Status verified 2015-11

CONDITIONS: Menorrhagia
MeSH Terms: conditions — Menorrhagia | interventions — Tranexamic Acid; Diosmin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tranexamic acid (Active Comparator)
  Interventions: Drug: Tranexamic Acid
- Diosmin (Active Comparator)
  Interventions: Drug: Diosmin

INTERVENTIONS:
Drug: Tranexamic Acid — use tranexamic acid oral tablets 500 mg two tablets every six hour with the onset of the first day of menstrual cycle till the end of bleeding then The amount of menstrual flow will be calculated by the PBAC
  Other Names: kapron
  Arms: Tranexamic acid
Drug: Diosmin — use diosmin oral tablets 500 mg t.d.s (three times daily) with the onset of the first day of menstrual cycle till the end of bleeding.then The amount of menstrual flow will be calculated by the PBAC
  Other Names: dycinon
  Arms: Diosmin

SUMMARY:
To compare the efficacy of tranexamic acid and diosmin in reducing menstrual blood loss in women having Intra Uterine Contraceptive Device (IUD) and suffer from menorrhagia.

ELIGIBILITY:
Inclusion Criteria:

* Women complaining from an menorrhagia secondary to a current copper IUD use.
* Age: 20-40years.
* Menorrhagia , will be defined as a PBAC-Score greater than 100.
* No systemic causes of abnormal uterine bleeding as hypertension and hemorrhagic blood diseases.
* No other local causes of abnormal uterine bleeding as, (fibroid, adenomyosis, polyps).
* No drugs decreasing blood coagulation.
* Well fitted IUD not misplaced.

Exclusion Criteria:

* Age <20y and >40y.
* Irregular menstrual cycle.
* Presence of systemic causes of abnormal uterine bleeding as hypertension and hemorrhagic blood diseases.
* Presence of other local causes of abnormal uterine bleeding as, (fibroid, adenomyosis, polyps).
* Taking drugs decrease blood coagulation.
* Misplaced IUD.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-09; Primary Completion 2016-01 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
The amount of reducing heavy menstrual flow will be calculated by the PBAC. | the first 24hours
  measure the bleeding rate will be by the pictorial blood assessment chart (PBAC).

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Alanwar, Cairo, Cairo Governorate, Egypt